CLINICAL TRIAL: NCT02945579
Title: Multicenter Trial for Eliminating Breast Cancer Surgery or Radiotherapy in Exceptional Responders to Neoadjuvant Systemic Therapy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016-0046; NCI-2016-01929 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2016-0046 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2016-10-24; First posted 2016-10-26 (Estimated); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Estrogen Receptor Negative; HER2 Positive Breast Carcinoma; HER2/Neu Negative; Invasive Breast Carcinoma; Progesterone Receptor Negative; Stage I Breast Cancer AJCC v7; Stage IA Breast Cancer AJCC v7; Stage IB Breast Cancer AJCC v7; Stage II Breast Cancer AJCC v6 and v7; Stage IIA Breast Cancer AJCC v6 and v7; Stage IIB Breast Cancer AJCC v6 and v7; Triple-Negative Breast Carcinoma
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Cohort A (Experimental): * Neoadjuvant chemotherapy therapy
  * Biopsy: if no disease remaining - stay on the study and receive radiation (skip breast surgery)
  * H&P and Imaging every 6 months
  Treatment (whole breast irradiation, EBRT) Within 12 weeks of completing neoadjuvant systemic therapy, patients undergo whole breast irradiation over 15-25 fractions on consecutive days. Patients then undergo EBRT boost over 7 fractions on consecutive days beginning the day following completion of whole breast irradiation.
  Interventions: Radiation: Undergo EBRT; Other: Laboratory Biomarker Analysis; Other: Quality-of-Life Assessment; Radiation: Partial Breast Irradiation
- Cohort B (Experimental): • Neoadjuvant endocrine therapy for 3 months
  Cohort B Radiation:
  Treatment (Stereotactic ablative radiotherapy -SABR) Following 3-6 months of endocrine therapy, if less than 25% tumor increase, patients undergo SABR irradiation over 5 fractions
  * Continued endocrine therapy for total of 5 years Biopsy 6-12months after radiation: if negative - additional endocrine therapy under the guidance of medical oncologist (skip breast surgery)
  * H&P and Imaging every 6 months
  Interventions: Radiation: Undergo EBRT; Other: Laboratory Biomarker Analysis; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Radiation: Partial Breast Irradiation
- Cohort C (Experimental): * Optional biopsy for nanomechanical biomarker assessment
  * Neoadjuvant chemotherapy therapy
  * Surgery (& optional biopsy nanomechanical biomarker assessment): if no disease remaining - stay on the study and skip radiation
  * H&P and Imaging every 6 months
  Interventions: Other: Laboratory Biomarker Analysis; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Cohort D (Experimental): * Optional biopsy for nanomechanical biomarker assessment
  * Chart review every year after surgery for 5 years
  * Eligible patients who have undergone the optional biopsy may later move to Cohort A or C if they meet all eligibility requirements and desire radiation omission.
  Interventions: Other: Questionnaire Administration

INTERVENTIONS:
Radiation: Undergo EBRT — Undergo EBRT
  Other Names: Definitive Radiation Therapy; SABR; External Beam Radiation Therapy; External Beam Radiotherapy; External Beam RT; external radiation; External Radiation Therapy; external-beam radiation
  Arms: Cohort A; Cohort B
Other: Laboratory Biomarker Analysis — Correlative studies
  Arms: Cohort A; Cohort B; Cohort C
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
  Arms: Cohort A; Cohort B; Cohort C
Other: Questionnaire Administration — Ancillary studies
  Arms: Cohort B; Cohort C; Cohort D
Radiation: Partial Breast Irradiation — Undergo partial breast irradiation
  Arms: Cohort A; Cohort B

SUMMARY:
This clinical trial studies eliminating surgery and/or radiation therapy in treating breast cancer patients. In HER2 positive and triple negative breast cancers, after systemic therapy, when image-guided biopsy shows no residual cancer, patients then receive standard breast radiotherapy with no surgery. In ER positive/HER2 negative breast cancers, after endocrine therapy and ablative radiotherapy, when image-guided biopsy shows no residual cancer, patients then receive standard endocrine therapy with no surgery. For patients who have HER2 positive and triple negative breast cancers and standard surgery, after systemic therapy, breast radiotherapy is being eliminated when the pathology from surgery shows no residual cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Cohort A1 and A2: To determine the 6 mo, 1, 2, 3, 5, 7, and 10 year biopsy confirmed ipsilateral breast tumor recurrence rate (IBTR, invasive and/or in situ) among patients who do not undergo surgery.

II. Cohort B: To determine the pCR rate 6 or 12 months after radiation therapy based on image-guided biopsy.

III. Cohort C: To determine the 6 mo, 1, 2, 3, 5, 7 and 10-year ipsilateral breast tumor recurrence rate among patients who undergo surgery alone without radiation.

SECONDARY OBJECTIVES:

I. Cohort B: To determine the 6 mo, 1, 2, 3, 5, 7 and 10--year biopsy confirmed ipsilateral breast tumor recurrence rate (IBTR, invasive and/or in situ) among patients who do not undergo surgery.

II. To determine the number (%) of patients where final biopsy reveals residual disease and quantify the residual disease (residual cancer burden, RCB) determined by routine pathologic examination of surgery specimens.

III. To assess baseline, 6 months, 1, 3, 5, 7, and 10 years decisional comfort of clinical trial participation using the Decisional Regret Scale (DRS).

IV. To determine patient-reported cosmetic outcome, breast pain, and functional status using the Breast Cancer Treatment Outcomes Scale (BCTOS) at baseline, 6 months, 1, 3, 5, 7, and 10 years.

V. To determine the 6 mo, 1, 2, 3, 5, 7, and 10 years incidence of ipsilateral breast and nodal recommendation and performance of biopsy based on breast imaging follow-up.

VI. Correlate "liquid biopsy" analyses (after standard routine NST, 6 months and one year post-radiotherapy or surgery) among protocol participants with pCR, utilizing circulating tumor cells (CTCs) and circulating tumor-DNA (ctDNA).

VII. Among patients who decide to proceed with routine surgery, record the results of final biopsy compared with routine pathologic examination of surgery specimens.

VIII. To determine patient-reported quality of life using the FACT B+4 instrument at baseline, 6 months, 1, 3, 5, 7, and 10 years after treatment.

IX. To explore if radiation genomic sensitivity scores and Oncotype performed on the initial diagnostic core biopsy specimen correlate with pCR rates in Cohort B.

X. To determine if changes in blood-based RNA Sequencing are elicited with radiation in Cohort B, measured at baseline, at the first 4-6 week follow-up after radiation, and at the 6 month post-radiation follow-up.

XI. In Cohort B to determine the 3-year rate of tumor control/ progression free survival (PFS).

XII. In Cohort C/D to determine whether nanomechanical biomarkers or quantification of stromal and tumor TILS can predict for low risk of local recurrence in exceptional responders who omit radiation therapy.

XIII. In Cohorts A/B/C/D: To record 6 mo, 1, 2, 3, 5, 7, and 10 year breast cancer disease-free and overall survival.

XIV. In Cohort D: Correlate nanomechanical biomarker analyses with pCR and/or local recurrence in patients with triple negative or her-2 positive breast cancer treated with lumpectomy +/- radiation.

OUTLINE:

For Cohorts A, within 12 weeks of completing neoadjuvant systemic therapy, patients undergo whole breast irradiation over 15-25 fractions on consecutive days. Patients then undergo external beam radiation therapy (EBRT) boost over 7 fractions on consecutive days beginning the day following completion of whole breast irradiation.

For Cohort B, patients will receive 3 months of neoadjuvant endocrine therapy, after which they will receive ablative partial breast irradiation over 5 fractions. Patients will then continue with endocrine therapy.

After completion of study treatment, patients are followed up every 6 months for 10 years.

ELIGIBILITY:
Inclusion Criteria:

* Cohort A1 and A2

  • Conditions for patient eligibility: Patients on this portion of the study can receive radiation treatment at any MD Anderson Cancer Center or any outside hospital and may be enrolled prior to, during, or following neoadjuvant systemic therapy provided they meet the following eligibility and ineligibility requirements noted below:
  1. Pathologically confirmed unicentric invasive breast cancer defined as radiologic clinical stage T1 or T2 (≤ 5 cm), N0 or N1 (≤ 4 abnormal axillary nodes on initial ultrasound), clinical stage M0.
  2. HER2 positive (IHC 3+ and or FISH amplified) or triple receptor negative (TN, ER/PR&amp;amp;amp;amp;amp;amp;amp;lt; 10% HER2 negative (IHC 1+ or 2+ FISH non-amplified) receiving any standard routine clinical NST regimen.
  3. Patient desires breast conserving therapy.
  4. Age 40 years or older. This age cutoff is justified because breast cancers in women under the age of 40 are known to have a significantly higher risk of IBTR presumably due to underlying biologic differences [124, 125].
  5. Female sex.
  6. If the patient has a history of a prior non-breast cancer, all treatment for this cancer must have been completed prior to study registration and the patient must have no evidence of disease for this prior non-breast cancer.
  7. Patient must have an initial nodal ultrasound that does not demonstrate more than four suspicious lymph nodes, any suspicious lymph nodes should be biopsied to determine if nodal metastatic disease present.
  8. Patient understands that the breast lesion size on final breast imaging must be less than or equal to 2 cm prior to the biopsy procedure being performed on study and if the biopsy shows residual carcinoma the patient will be taken off study.
* Cohort B1 and B2

  • Conditions for patient eligibility: Patients on this portion of the study will be limited to receive radiation treatment at MD Anderson Cancer Center or other approved locations and must be enrolled prior to any neoadjuvant systemic therapy provided they meet the following eligibility and ineligibility requirements noted below:
  1. ER and/or PR positive, HER2 negative
  2. Clinical stage T1N0M0, unicentric non-lobular breast cancer, no lymphovascular space invasion,
  3. At least 40 years of age.
  4. Oncotype ≤ 25 if age ≥ 50 years
  5. Oncotype 0-20 and tumor size ≤ 1.5cm if age 40-49 years.
  6. Patient agrees to take anti-estrogen therapy and is interested in breast conservation
  7. Female sex.
  8. If the patient has a history of a prior non-breast cancer, all treatment for this cancer must have been completed prior to study registration and the patient must have no evidence of disease for this prior non-breast cancer.
  9. No history of prior radiation to the area of the breast that would require protocol-mandated treatment
* Cohort C

  • Conditions for patient eligibility: Patients on this portion of the study can receive surgical treatment at any MD Anderson Cancer Center or any outside hospital and may be enrolled prior to or following neoadjuvant systemic therapy provided they meet the following eligibility and ineligibility requirements noted below:
  1. Pathologically confirmed invasive breast cancer defined as radiologic clinical stage T1 or T2 (≤ 5 cm), N0, clinical stage M0 and HER2 positive (IHC 3+ and or FISH amplified) receiving any standard routine clinical NST regimen containing her-2 directed therapy OR Pathologically confirmed invasive breast cancer defined as radiologic clinical stage T1 (≤ 2 cm), N0, clinical stage M0 and triple negative, receiving any standard routine clinical NST regimen.
  2. For cohort C patients participating in the optional pretreatment biopsy, the patient should be able undergo biopsy or surgery of the primary tumor site of suspected or proven invasive breast cancer and should be planned to receive neoadjuvant systemic therapy.
  3. Patient desires breast conserving therapy.
  4. Age 30 years or older if HER2 positive. Age 50 or older if HER2 negative (triple negative).
  5. Female sex.
  6. If the patient has a history of a prior non-breast cancer, all treatment for this cancer must have been completed prior to study registration and the patient must have no evidence of disease for this prior non-breast cancer.
  7. Patient must have an initial nodal ultrasound that does not demonstrate suspicious lymph nodes; any suspicious lymph nodes should be biopsied to determine if nodal metastatic disease present.
  8. Patient must have no evidence of residual invasive tumor or DCIS on pathologic review of the lumpectomy surgical specimen
  9. Patient must have no evidence of metastatic disease or isolated tumor cells involving the lymph nodes on pathologic review of the lymph node surgical specimen. If treatment effect in the nodes is noted on the pathology report, the investigators would generally discourage enrollment on this protocol.
  10. Unifocal disease or limited multifocal disease that can be excised in a single lumpectomy specimen
* Cohort D (MD Anderson Houston patients only)

  * Conditions for patient eligibility: Patients on this portion of the study meet all eligibility requirements for cohort C, but have not enrolled onto the study to omit radiation. Patients in Cohort D can be identified at the time of diagnosis or prior to lumpectomy. They are not required to participate in one of the treatment arms of the study, but can ultimately choose to move to an omission Cohort at a later time point.

3.5.1 Patients with triple negative or her-2 positive tumor who are amenable to breast conserving treatment and have received or are planned for neoadjuvant systemic therapy prior to surgery are eligible for Cohort D.

3.5.2 Eligible patients in cohort D who have undergone optional ARTIDIS biopsies of the primary breast tumor at the time of diagnosis, prior to starting neoadjuvant therapy, or following completion of systemic therapy, at the time of surgery, may later move to Cohort A or C if they meet all eligibility requirements and ultimately desire surgery or radiation omission

Exclusion Criteria:

1. Radiologic evidence for a stage T3 or clinical stage T4 breast cancer in Cohort A1/A2/C; radiologic evidence for a stage T2-T3 or clinical stage T4 breast cancer in Cohort B1/B2.
2. Clinical or pathologic evidence for distant metastases.
3. Prior diagnosis of invasive or ductal carcinoma in situ breast cancer in the ipsilateral breast.
4. Clinical evidence of progression of disease &amp;amp;amp;amp;amp;amp;amp;gt;20% in the breast or new evidence of nodal metastases.
5. Patient is known to be pregnant.
6. Patient is participating in a NST protocol in which surgical excision of the breast and or lymph nodes are required in Cohort A1/A2/B1/B2.

Min Age: 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2017-01-20 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Ipsilateral breast tumor recurrence-free survival (IBT-RFS) | From confirmation of pathologic complete response (pCR) to the time of ipsilateral breast tumor recurrence or death, whichever occurs first or the time of last contact, assessed for up to 10 years
  Will monitor IBT-RFS using the method of Thall et al. Will be estimated using the Kaplan-Meier method log-rank test will be performed to test the difference in time-to-event distributions between patient groups. Cox proportional hazards model will be used to include multiple covariates in the time-to-event analysis.
Overall survival | Up to 10 years
  Will be estimated using the Kaplan-Meier method log-rank test will be performed to test the difference in time-to-event distributions between patient groups. Cox proportional hazards model will be used to include multiple covariates in the time-to-event analysis.

OTHER OUTCOMES:
Change in biomarkers in blood and plasma | 3 months, 3-8 weeks post radiation therapy (if applicable), 6 months, 12 months]
  Biomarkers in blood and plasma, specifically CTC and cDNA, will be assessed by exploratory data analysis and graphical methods, which will be applied to examine distributions and to identify data errors and outliers. Linear mixed effect models for repeated measures analysis will be employed to assess the change of the data over time with multi-covariates including disease characteristics (tumor stage, site, pathology), and other patient prognostic factors.
Residual cancer burden (RCB) | Up to 10 years
  Will be assessed by biopsy and routine surgery. Descriptive statistics will be used. The final biopsy will be compared with the response status determined by routine pathologic examination of surgery specimens using McNemar test.
Incidence of ipsilateral breast and nodal recommendation and performance of biopsy based on breast imaging follow-up | Up to 10 years
  Multivariable logistic regression analysis using generalized estimating equations to take the intra-patient correlation into account will be used to determine factors significantly associated with the outcome.
Quality of Life measured by DRS questionnaire | Baseline, 6 months, 12 months, 36 months, 60 months, 84 months, and 120 months]
  The Decisional Regret Scale (DRS) questionnaire will assess the decisional comfort of the clinical trial participant.
  Question answers range : Strongly Agree, Agree, Neither Agree Nor Disagree, Disagree, or Strongly Agree
Quality of Life measured by BCTOS questionnaire | Baseline, 6 months, 12 months, 36 months, 60 months, 84 months, and 120 months]
  The Breast Cancer Treatment Outcome Scale (BCTOS) will assess patient-reported cosmetic outcome, breast pain, and functional status by comparing the affected breast with her unaffected breast.
Quality of Life measured by FACT-B+4 questionnaire | Baseline, 6 months, 12 months, 36 months, 60 months, 84 months, and 120 months]
  The FACT-B+4 will assess the general quality of life of the patient.

CONTACTS AND LOCATIONS:
Overall Officials: Henry M Kuerer, Principal Investigator — M.D. Anderson Cancer Center
Locations (8):
- United States (8):
  - MD Anderson Cancer Center - Banner, Gilbert, Arizona
  - Baptist MD Anderson Cancer Center, Jacksonville, Florida
  - Queen's Medical Center, Honolulu, Hawaii
  - Mayo Clinic, Rochester, Minnesota
  - Cooper Hospital Univ Med Ctr, MD Anderson at Cooper Voorhees, Voorhees Township, New Jersey
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - M D Anderson Cancer Center, Houston, Texas

REFERENCES:
- [Derived] Kuerer HM, Valero V, Smith BD, Krishnamurthy S, Diego EJ, Johnson HM, Lin H, Shen Y, Lucci A, Shaitelman SF, Mitchell MP, Boughey JC, White RL, Hunt KK, Yang WT, Rauch GM; Exceptional Responders Study Group. Selective Elimination of Breast Surgery for Invasive Breast Cancer: A Nonrandomized Clinical Trial. JAMA Oncol. 2025 May 1;11(5):529-534. doi: 10.1001/jamaoncol.2025.0207. PMID 40152443
- [Derived] Johnson HM, Lin H, Shen Y, Diego EJ, Krishnamurthy S, Yang WT, Smith BD, Valero V, Lucci A, Sun SX, Shaitelman SF, Mitchell MP, Boughey JC, White RL, Rauch GM, Kuerer HM; Exceptional Responders Study Group. Patient-Reported Outcomes of Omission of Breast Surgery Following Neoadjuvant Systemic Therapy: A Nonrandomized Clinical Trial. JAMA Netw Open. 2023 Sep 5;6(9):e2333933. doi: 10.1001/jamanetworkopen.2023.33933. PMID 37707811
- [Derived] Kuerer HM, Smith BD, Krishnamurthy S, Yang WT, Valero V, Shen Y, Lin H, Lucci A, Boughey JC, White RL, Diego EJ, Rauch GM; Exceptional Responders Clinical Trials Group. Eliminating breast surgery for invasive breast cancer in exceptional responders to neoadjuvant systemic therapy: a multicentre, single-arm, phase 2 trial. Lancet Oncol. 2022 Dec;23(12):1517-1524. doi: 10.1016/S1470-2045(22)00613-1. Epub 2022 Oct 25. PMID 36306810
- [Derived] Hariharan N, Rao TS, Rajappa S, Naidu CCK. Precision medicine - A new era in multidisciplinary care. Cancer Treat Res Commun. 2022;32:100577. doi: 10.1016/j.ctarc.2022.100577. Epub 2022 May 17. No abstract available. PMID 35617923
- See also: MD Anderson Cancer Center — http://www.mdanderson.org

DOCUMENTS (1):
  • Informed Consent Form (2024-12-16): https://cdn.clinicaltrials.gov/large-docs/79/NCT02945579/ICF_000.pdf